CLINICAL TRIAL: NCT04450485
Title: Does Mini Mid-Vastus Approach Have An Advantageous Effect On Rapid Recovery Protocols Over Medial Parapatellar Approach In Total Knee Arthroplasty? A Prospective, Randomized, Single-Blinded Study
Brief Title: Surgical Approach in Fast Track Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Harun Resit Gungor, MD, Associated Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018TIPF017
Record Dates: First submitted 2020-06-23; First posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Knee Arthroplasty, Total
Keywords: Total knee arthroplasty; Surgical approach; Fast track
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: Patients planned for fast track protocol applied total knee arthroplasty randomized into two groups by a computer program to generate random numbers and assign participants to either to mini mid-vastus or medial para-patellar surgical approach group
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and outcomes assessor are blinded to the type of surgical approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medial para-patellar approach (Active Comparator): Fast track protocol applied total knee arthroplasty patients operated by using medial para-patellar approach
  Interventions: Procedure: Total knee arthroplasty
- Mini mid-vastus approach (Active Comparator): Fast track protocol applied total knee arthroplasty patients operated by using mini mid-vastus approach
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — Total knee arthroplasty

SUMMARY:
Nowadays, due to the demands to improve life and health conditions of osteoarthritis patients, more effective surgical treatment methods are needed to obtain satisfactory results when performing total knee arthroplasty (TKA). Fast-track surgical protocols are evidence based multidisciplinary approaches targeted on multimodal patient care and primarily focused on enhancing rapid functional recovery of the patients. These protocols recommend use of minimal invasive approaches for TKA patients to enhance rapid recovery. Although studies in the literature has been reported similar results in medial para-patellar approach (MPP) and minimal invasive approaches in long terms, better surgical outcomes in short term in favor of minimal invasive approaches also encouraged fast-track protocol builders to prefer minimal invasive approaches. However, this recommendation is not evidence based and there is no study comparing surgical outcomes between minimal invasive approaches and MPP approach in terms of pain, length of hospital stays and functional recovery in fast-track TKA patients. Therefore, we aimed to compare the effects of mini mid-vastus (MMV) and MPP approaches on postoperative clinical results (pain, quality of life, functional outcome, and length of hospital stay) in fast-track TKA patients, and to decide whether any additional achievements are obtained with MMV approach in this patient group.

DETAILED DESCRIPTION:
Nowadays, due to the demands to improve life and health conditions of OA patients, more effective surgical treatment methods are needed to obtain satisfactory results when performing total knee arthroplasty (TKA). Fast-track surgical protocols are evidence based multidisciplinary approaches targeted on multimodal patient care and primarily focused on enhancing rapid functional recovery of the patients. These protocols include patient education to cope with anxiety and stress of surgery, nutritional planning and avoidance of long hours of fasting, preemptive analgesia, avoidance of tourniquet use, rational antibiotic prophylaxis, local infiltration anesthesia, and early physical therapy modalities. The ultimate aims of assembling these surgical protocols are to decrease mortality and morbidity, length of hospital stay, and eventually hospital costs while obtaining maximum patient satisfaction.

Surgical approaches when performing TKA operations includes standard medial parapatellar (MPP) approach and minimal invasive approaches such as mini midvastus (MMV) and subvastus (SV) approaches. Possible advantages of not performing quadriceps tendon splitting in MV surgical approach (such as less pain, earlier functional recovery, enhanced quadriceps muscle strength, and better ROM) convinced surgeons to prefer minimal invasive approaches to MPP approach when performing rapid recovery protocols in TKA patients. In addition, better surgical outcomes with traditional protocols in short term reports in favor of minimal invasive approaches also encouraged fast-track protocol builders to prefer minimal invasive approaches. However, these recommendations are not evidence based and, to our knowledge, there is no study comparing surgical outcomes between minimal invasive approaches and MPP approach in terms of pain, length of hospital stay and functional recovery in fast-track TKA patients. Therefore, we aimed to compare the effects of MMV and MPP approaches on postoperative clinical results (pain, quality of life, functional outcome, and length of hospital stay) in fast-track TKA patients, and to decide whether any additional achievements are obtained with MMV approach in this patient group. Our secondary outcome measures were length of operation time, blood loss and postoperative component alignments.

Clinical and demographic variables of the participants were recorded and patients were evaluated preoperatively, at postoperative fourth and twelfth week by a blinded observer. Knee range of motion was assessed with digital goniometer (HALO Medical Devices, Australia); quadriceps muscle strength was measured (unit=newton(N)) with hand-held dynamometer (Commander Muscle Tester, J Tech, USA); The Western Ontario and McMaster Universities Arthritis Index (WOMAC) and Knee injury and Osteoarthritis Outcome Score (KOOS) was used to determine patient-reported activity limitations; 30-sec chair-stand test and stair-climb test were performed for performance-based activity limitations; Short Form-36 (SF-36) was used for quality of life evaluations.

Alignment analysis Long leg radiographs of the patients were evaluated preoperatively and postoperatively by using a digital orthopedic templating software-Materialise OrthoView (OrthoView version 7, Materialise HQ, Technologielaan 15 3001 Leuven, Belgium). Hip-knee-ankle angles (HKA), femorotibial angles, lateral proximal femoral angles (LPFA), lateral distal femoral angles (LDFA), medial proximal tibial angles (MPTA), lateral distal tibial angles (LDTA), tibial posterior slope angles were all measured and recorded by a blinded observer.

Preoperative patient education classes All the patients were received preoperative informative classes about TKA procedure, nutritional and nursing support, physical therapy and rehabilitation applications. Booklets concerning all these classes were also handed out to all patients.

Anesthesia Protocol Excluding diabetics, all the patients were received oral carbohydrate (%12.5 carbohydrate liquid solution-Fantomalt, Nutricia) loading on the night before the operation (between 19:00 and 23:00) and 2 hours before the operation. Solid foods were allowed up to 6 hours before the operation and liquids allowed up to 2 hours preoperatively. Early oral feeding was started at 4 to 6 hours postoperatively for all patients. Intravenous midazolam 1-2 mg and fentanyl 50-100 μg were applied to all patients 30-45 minutes preoperatively. Except 12 patients, all patients received spinal anesthesia. Seven patients due to previous lumber fusion and 5 patients due to personal preference were received general anesthesia.

Surgical Technique All the operations were performed by the same surgeon using the same brand and type of prosthesis. MPP and MMV approaches were performed as described in the literature. All the patients received posterior stabilized fixed bearing TKA (NexGen Legacy® Posterior Stabilized Knee-Fixed Bearing, Zimmer-Biomet Inc., Warsaw, Indiana 46580, ABD), and high viscosity polymethyl methacrylate (PMMA) bone cement (Oliga-G21 srl-Vias. Pertini, 8-41039 San Posidonia (MO)-Italy). All the operations were performed without using tourniquet.

Local infiltration anesthesia (LIA) (20 cc bupivacaine hydrochloride, 1 gr fentanyl, 1 gr cefazolin sodium, 0.3 ml epinephrine, and dilute volume of physiologic serum (%0,9 NaCl) to 50 cc) to posterior capsule just before the application of permanent implants, and to anterior capsule, prepatellar fat pad and peri ligamentous nociceptive receptors following consolidation of bone cement was injected.

One gram of tranexamic acid was injected intravenously (iv) at least 30 minutes before the incision, 1 gr diluted to 30 cc by physiologic serum (%0,9 NaCl) was given intraarticularly following the closure of the wound, and another 1 gr was infused 2 hours after the operation.

Preoperative and postoperative analgesia protocol For preemptive analgesia, paracetamol 500 mg tablets were prescribed 3 times 2 tablets per day beginning from 3 days before the operation. One gram of iv infusion of paracetamol was given just after the operation in postoperative care unit and continued as 3 times 1gr iv infusion. First line rescue analgesic was intramuscular 75 mg diclofenac sodium and second line analgesic was iv 100 mg tramadol hydrochloride.

Antibiotic and thrombosis prophylaxis protocol One gr of cefazolin sodium iv was applied 30 minutes before the incision as antibiotic prophylaxis. Low molecular weight heparin-enoxaparin sodium 4000 iu/0.8 ml/day was used subcutaneously as thromboembolic prophylaxis starting at the 6-8 hours postoperatively and continued for 20 days.

Rehabilitation protocol and discharge criteria The patients were mobilized at the 4th hour following surgery and standard physiotherapy program was scheduled during hospitalization (cold-pack -once in every 2 hours for 15 minutes, ankle pump exercises, quadriceps isometric exercises, active assisted heel slide exercises in bed and knee flexion exercises in sitting position/3 sets×10 repeats). The patients were evaluated regularly every two hours during postoperative period and those fulfilling discharge criteria were released from the hospital and length of hospital stay was recorded for every patient. The standard discharge criteria were as follows: VAS score at rest <3, VAS score during mobilization <5, able to get dressed independently, able to get in and out of bed, able to sit and rise from a chair/toilet seat, independence in personal care, mobilization with walker/crutches, able to walk >70 meters without risk of fall with walking aid, no incision problem.

The discharged patients were instructed for a standard home-based exercise program. Patients were also asked to visit the ward at a biweekly interval for the update of the exercise program for the first 8 weeks. 15-40 minutes of walking exercises were also prescribed for 5 days/week between 9th and 12th weeks.

Statistical analysis Priori power analysis concerning quadriceps muscle strength showed that at an effect size of d=0.7, 52 patients are needed (26 patients for each group) to obtain 80 % power (1-beta=0.80) with 95 % confidence interval (alpha=0.05).

The data was analyzed using SPSS 24.0 (IBM Corp. Released 2016. IBM SPSS Statistics for Windows, Version 24.0. Armonk, NY: IBM Corp.) package program. Continuous variables were given as mean ± standard deviation, median (minimum and maximum) and categorical variable values were presented as absolute numbers and percentages. The conformity of continuous variables with normal distribution was evaluated using the Shapiro-Wilk test. Independent Samples t-test for parametric test assumptions and Mann-Whitney U Test for non-parametric test assumptions were used for comparison of the groups. One-way repeated-measure ANOVA was used to compare the normally distributed data from the parameters repeatedly measured in the inner-group analysis, and Friedman analysis of variance was performed for the remaining data set. Statistical significance was set at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for unilateral TKA surgery due to primary OA
* Patients capable of understanding verbal and written instructions.

Exclusion Criteria:

* Revision TKA surgery
* ASA score >3
* previous major orthopedic surgery in either lower extremities
* neurologic compromise
* psychiatric problems
* regular hypnotic and/or anxiolytic medication usage
* dementia
* patients participated in a particular physical activity program within the last 3 months.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Pain preoperative | Baseline (preoperatively)
  Visual Analog Scale used to assess pain
Pain postoperative 1 | at postoperative fourth weeks
  Visual Analog Scale used to assess pain
Pain postoperative 2 | at postoperative twelfth weeks
  Visual Analog Scale used to assess pain
Knee Range of Motion preoperative | Baseline (preoperatively)
  Digital goniometer (HALO Medical Devices, Australia) used to assess knee range of motion
Knee Range of Motion postoperative 1 | at postoperative fourth week
  Digital goniometer (HALO Medical Devices, Australia) used to assess knee range of motion
Knee Range of Motion postoperative 2 | at postoperative twelfth week
  Digital goniometer (HALO Medical Devices, Australia) used to assess knee range of motion
Quadriceps muscle strength preoperative | Baseline (preoperatively)
  Quadriceps muscle strength is measured (unit=newton(N)) with hand-held dynamometer (Commander Muscle Tester, J Tech, USA)
Quadriceps muscle strength postoperative 1 | at postoperative fourth weeks
  Quadriceps muscle strength is measured (unit=newton(N)) with hand-held dynamometer (Commander Muscle Tester, J Tech, USA)
Quadriceps muscle strength postoperative 2 | at postoperative twelfth weeks
  Quadriceps muscle strength is measured (unit=newton(N)) with hand-held dynamometer (Commander Muscle Tester, J Tech, USA)
Patient-reported activity limitations preoperative | Baseline (preoperatively)
  The Western Ontario and McMaster Universities Arthritis Index and Knee injury and Osteoarthritis Outcome Score are used
Patient-reported activity limitations postoperative 1 | at postoperative fourth weeks
  The Western Ontario and McMaster Universities Arthritis Index and Knee injury and Osteoarthritis Outcome Score are used
Patient-reported activity limitations postoperative 2 | at postoperative twelfth weeks
  The Western Ontario and McMaster Universities Arthritis Index and Knee injury and Osteoarthritis Outcome Score are used
Performance-based activity limitations-preoperative | Baseline (preoperatively)
  30-sec chair-stand test and stair-climb test are used
Performance-based activity limitations- postoperative 1 | at postoperative fourth weeks
  30-sec chair-stand test and stair-climb test are used
Performance-based activity limitations - postoperative 2 | at postoperative twelfth weeks
  30-sec chair-stand test and stair-climb test are used
Quality of life-preoperative | Baseline (preoperatively)
  Short Form-36 (SF-36) is used
Quality of life-preoperative- postoperative 1 | at postoperative fourth weeks
  Short Form-36 (SF-36) is used
Quality of life-preoperative- postoperative 2 | at postoperative twelfth weeks
  Short Form-36 (SF-36) is used
Length of hospital stay | through study completion, an average of 1 year
  Length of hospital stay is measured beginning from the hospitalization of the patient and ending at discharge of the patients (unit-hours)

SECONDARY OUTCOMES:
Length of operation time | the surgery
  Length of operation time is measured in minutes during the surgery
Amount of blood loss | through study completion, an average of 1 year
  Amount of blood loss is measured from the suction drainage (unit-milliliters)
postoperative component alignments | through study completion, an average of 1 year
  Long leg radiographs of the patients are evaluated postoperatively by using a digital orthopedic templating software-Materialise OrthoView (OrthoView version 7, Materialise HQ, Technologielaan 15 3001 Leuven, Belgium).

CONTACTS AND LOCATIONS:
Overall Officials: Harun R Gungor, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University Medical Faculty, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Husted H. Fast-track hip and knee arthroplasty: clinical and organizational aspects. Acta Orthop Suppl. 2012 Oct;83(346):1-39. doi: 10.3109/17453674.2012.700593. PMID 23205862
- [Background] Stowers MD, Manuopangai L, Hill AG, Gray JR, Coleman B, Munro JT. Enhanced Recovery After Surgery in elective hip and knee arthroplasty reduces length of hospital stay. ANZ J Surg. 2016 Jun;86(6):475-9. doi: 10.1111/ans.13538. Epub 2016 Mar 28. PMID 27018137
- [Background] Heekin RD, Fokin AA. Mini-midvastus versus mini-medial parapatellar approach for minimally invasive total knee arthroplasty: outcomes pendulum is at equilibrium. J Arthroplasty. 2014 Feb;29(2):339-42. doi: 10.1016/j.arth.2013.05.016. Epub 2013 Jun 19. PMID 23790343
- [Background] Karpman RR, Smith HL. Comparison of the early results of minimally invasive vs standard approaches to total knee arthroplasty: a prospective, randomized study. J Arthroplasty. 2009 Aug;24(5):681-8. doi: 10.1016/j.arth.2008.03.011. Epub 2008 Jun 6. PMID 18538536
- [Background] Chin PL, Foo LS, Yang KY, Yeo SJ, Lo NN. Randomized controlled trial comparing the radiologic outcomes of conventional and minimally invasive techniques for total knee arthroplasty. J Arthroplasty. 2007 Sep;22(6):800-6. doi: 10.1016/j.arth.2006.10.009. Epub 2007 Apr 20. PMID 17826268
- [Background] Dalury DF, Jiranek WA. A comparison of the midvastus and paramedian approaches for total knee arthroplasty. J Arthroplasty. 1999 Jan;14(1):33-7. doi: 10.1016/s0883-5403(99)90199-7. PMID 9926950
- [Background] White RE Jr, Allman JK, Trauger JA, Dales BH. Clinical comparison of the midvastus and medial parapatellar surgical approaches. Clin Orthop Relat Res. 1999 Oct;(367):117-22. PMID 10546605
- [Background] Stevens-Lapsley JE, Bade MJ, Shulman BC, Kohrt WM, Dayton MR. Minimally invasive total knee arthroplasty improves early knee strength but not functional performance: a randomized controlled trial. J Arthroplasty. 2012 Dec;27(10):1812-1819.e2. doi: 10.1016/j.arth.2012.02.016. Epub 2012 Mar 28. PMID 22459124
- [Background] Lin WP, Lin J, Horng LC, Chang SM, Jiang CC. Quadriceps-sparing, minimal-incision total knee arthroplasty: a comparative study. J Arthroplasty. 2009 Oct;24(7):1024-32. doi: 10.1016/j.arth.2008.07.005. Epub 2008 Aug 30. PMID 18757172
- [Background] Nestor BJ, Toulson CE, Backus SI, Lyman SL, Foote KL, Windsor RE. Mini-midvastus vs standard medial parapatellar approach: a prospective, randomized, double-blinded study in patients undergoing bilateral total knee arthroplasty. J Arthroplasty. 2010 Sep;25(6 Suppl):5-11, 11.e1. doi: 10.1016/j.arth.2010.04.003. Epub 2010 Jun 11. PMID 20541889
- [Background] Kazarian GS, Siow MY, Chen AF, Deirmengian CA. Comparison of Quadriceps-Sparing and Medial Parapatellar Approaches in Total Knee Arthroplasty: A Meta-Analysis of Randomized Controlled Trials. J Arthroplasty. 2018 Jan;33(1):277-283. doi: 10.1016/j.arth.2017.08.025. Epub 2017 Aug 30. PMID 28947369